CLINICAL TRIAL: NCT03548948
Title: Obesity, Iron Regulation and Colorectal Cancer Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Principal Investigator, Lisa Tussing-Humphreys, Associate Professor, University of Illinois at Chicago
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2014-0721
Record Dates: First submitted 2018-05-07; First posted 2018-06-07 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Colon Inflammation; Iron Malabsorption; Obesity; Diet Modification
MeSH Terms: conditions — Colitis; Obesity

STUDY DESIGN:
Intervention Model Description: 1. Typical American Diet with "high" heme/non-heme iron (16 mg)
  2. Typical American Diet with "low" iron (8 mg)
  3. Plant-based Diet with "high" non-heme iron (16 mg)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High heme iron diet (Other)
  Interventions: Other: High heme iron diet
- Low iron diet (Other)
  Interventions: Other: Low iron diet
- Plant-based high non-heme iron diet (Other)
  Interventions: Other: Plant-based high non-heme iron diet

INTERVENTIONS:
Other: High heme iron diet — A "Typical American" diet with "high" heme/non-heme iron" (18 mg total). Diet is isocaloric and has a macronutrient composition of total fat 35%, carbohydrates 50%, protein 15% of calories and fiber 9g/1000 calories. Subjects consumes the diet for 3 weeks with a minimum 3 week washout before the next diet.
  Arms: High heme iron diet
Other: Low iron diet — A "Typical American" diet with "low" heme/non-heme iron" (8 mg total). Diet is isocaloric and has a macronutrient composition of total fat 35%, carbohydrates 50%, protein 15% of calories and fiber 9g/1000 calories. Subjects consumes the diet for 3 weeks with a minimum 3 week washout before the next diet.
  Arms: Low iron diet
Other: Plant-based high non-heme iron diet — A plant-based diet with "high" non-heme iron" (18 mg total). Diet is isocaloric and has a macronutrient composition of total fat 35%, carbohydrates 50%, protein 15% of calories and fiber 9g/1000 calories. Subjects consumes the diet for 3 weeks with a minimum 3 week washout before the next diet.
  Arms: Plant-based high non-heme iron diet

SUMMARY:
Obesity is an independent risk factor for colorectal cancer (CRC) although the underlying mechanisms have not been elucidated. Dietary nutrients play a key role in both the prevention and promotion of CRC. While iron is an essential nutrient, excess iron is associated with carcinogenesis. Unlike the systemic compartment, the intestinal lumen lacks an efficient system to regulate iron. In conditions when dietary iron malabsorption and intestinal inflammation co-exist, greater luminal iron is associated with increased intestinal inflammation and a shift in the gut microbiota to more pro-inflammatory strains. However, treatments designed to reduce luminal, including diet restriction and chelation, are associated with lower intestinal inflammation and the colonization of protective gut microbes. Obesity is associated with inflammation-induced, hepcidin-mediated, iron metabolism dysfunction characterized by iron deficiency and dietary iron malabsorption. Obesity is also linked to intestinal inflammation. Currently, there is a fundamental gap in understanding how altered iron metabolism impacts CRC risk in obesity.

The investigator's objective is to conduct a crossover controlled feeding trial of: 1) a "Typical American" diet with "high" heme/non-heme iron", 2) a "Typical American" diet with "low" iron, and 3) a Mediterranean diet with "high" non heme iron and examine effects on colonic and systemic inflammation and the gut microbiome.

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as Hispanic, African American, or Caucasian.
* Meet body mass index (BMI > = 30.0 kg/m2) and C-reactive protein (CRP) criteria (> 2.0 mg/dl)
* Post-menopausal (no menstruation in the past 12 months)
* Weight stable (< 3% weight change in the past 3 months)
* Non-smoker
* No major medical problems
* Have a working phone
* No known allergies, intolerance, medical, secular or religious dietary restrictions

Exclusion Criteria:

* Chronic constipation (less than three stools per week for several months)
* History or intestinal cancer, inflammatory bowel disease, celiac disease, or malabsorptive bariatric surgery
* Previous intestinal surgery
* H pylori infection or taking H2 blockers (e.g., Zantac, Pepcid) /antacids (e.g., Rolaids) more than 3 times per week
* Significant blood loss or blood donation in past 3 months
* Active gastrointestinal bleed
* Any surgery in the past 3 months
* Hemochromatosis
* Sickle cell disease
* Hereditary polyposis
* Rheumatoid arthritis
* Type I or Type II diabetes
* Smoker
* Antibiotic use in the past 2 months
* Excessive alcohol consumption [> 2 standard alcoholic drinks (12 ounces of beer, 5 ounces of wine, 1 shot of hard liquor) per day]
* Aspirin use >81 mg/day OR >325 mg/every other day
* Regularly taking probiotics, fiber supplements, Orlistat (over the counter brand name: Alli), or steroids (inhaled or oral)

Ages: 55 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2015-07-15 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Change in colonic inflammation | Baseline and post-diet (day 22) for each of the three 3-week diets
  Fecal calprotectin, a proxy for colon tissue inflammation, will be measured from stool an calprotectin immunoassay

SECONDARY OUTCOMES:
Change in systemic inflammation | Baseline and post-diet (day 22) for each of the three 3-week diets
  Circulating C-reactive protein, Interleukin-6 (IL-6) and Tumor necrosis factor-alpha (TNF-a) will be measured from serum using immunoassays.
Change in stool microbial community profile at the phylum and genus level | Baseline and post-diet (day 22) for each of the three 3-week diets
  Stool samples to analyze the composition of the microbiota, extracted bacterial genomic DNA will be used as a template for polymerase chain reactions targeting the V4 variable regions of the 16S ribosomal ribonucleic acid gene. Amplicons generated from polymerase chain reaction will be run on the Illumina MiSeq sequencing platform to profile microbial communities at the phylum and genus level.
Change in serum hepcidin | Baseline and post-diet (day 22) for each of the three 3-week diets
  Serum hepcidin will be measured using an immunoassay

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Tussing-Humphreys, PhD, MS, RD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States